CLINICAL TRIAL: NCT00000655
Title: A Randomized, Double-Blind Study of 566C80 Versus Septra (Trimethoprim/Sulfamethoxazole) for the Treatment of Pneumocystis Carinii Pneumonia in AIDS Patients
Brief Title: A Randomized, Double-Blind Study of 566C80 Versus Septra (Sulfamethoxazole/Trimethoprim) for the Treatment of Pneumocystis Carinii Pneumonia in AIDS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 167; NIAID 90-CC-185; Protocol #03; FDA 53A; Project P71
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Naphthoquinones; Antifungal Agents; Acquired Immunodeficiency Syndrome; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Atovaquone; Trimethoprim, Sulfamethoxazole Drug Combination

INTERVENTIONS:
Drug: Atovaquone
Drug: Sulfamethoxazole-Trimethoprim

SUMMARY:
To evaluate the effectiveness of atovaquone (566C80) compared to a standard antipneumocystis agent, (SMX/TMP), for the treatment of mild to moderate Pneumocystis carinii pneumonia (PCP) in AIDS patients. To compare the safety of short-term (21 days) treatment with 566C80 and SMX/TMP in AIDS patients with an acute episode of PCP.

Standard therapies for acute treatment of PCP involve either SMX/TMP or pentamidine isetionate. Although both treatments are equally effective, side effects prevent completion of therapy in 11-55 percent of patients.

DETAILED DESCRIPTION:
Standard therapies for acute treatment of PCP involve either SMX/TMP or pentamidine isetionate. Although both treatments are equally effective, side effects prevent completion of therapy in 11-55 percent of patients.

Patients are randomized into one of two treatment groups to receive either (1) 566C80 for 21 days, or (2) SMX/TMP for 21 days. Patients will be stratified according to severity of PCP. Group A will be those with an arterial-alveolar (A-a) DO2 < 35 mm Hg. Group B will have an A-a DO2 of 35-45 mm Hg., and will also be required to receive therapy with Corticosteroids. All doses are taken with food. During the 21 days of treatment, patients are examined clinically for adverse effects and have hematology (blood-related) and clinical chemistry studies conducted a minimum of 2 times weekly. More frequent monitoring may be required at the discretion of the investigator. To evaluate the effectiveness of study medication, the clinical status of each patient is evaluated 2 to 3 times per week (e.g., dyspnea score, cough score, chest tightness/pain score, vital signs). Also, on days 7 and 21 of treatment, an arterial blood gas measurement and chest X-ray are performed. Patients who experience severe toxicities will be discontinued from the study and placed on alternative therapy. Patients will also be removed from study if they show significant clinical deterioration within the first 7 days of therapy or if there is no improvement after 10 days of therapy. This study involves a double placebo with one group randomized to receive oral 566C80 and placebo tablets which look like SMX/TMP while the other group will receive SMX/TMP and placebo tablets looking like 566C80.

ELIGIBILITY:
Inclusion Criteria

Patient must have the following:

* Presumptive diagnosis of AIDS as defined by the CDC.
* Untreated Pneumocystis carinii pneumonia (PCP).
* Willingness and ability to give informed consent.

Prior Medication:

Allowed:

* Prophylactic therapy for Pneumocystis carinii pneumonia (PCP) including aerosolized pentamidine or sulfamethoxazole/trimethoprim (SMX/TMP) (at a dose no greater than two DS tablets twice daily).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Judged by the investigator to be in impending respiratory failure.
* Malabsorption or vomiting that would, in the judgment of investigator, potentially limit the retention and absorption of an oral therapy.
* Concurrent bacterial, fungal, or viral pneumonitis, pulmonary Kaposi's sarcoma or other concurrent illness, or chronic pulmonary disease that, in the investigator's opinion, would make interpretation of drug efficacy difficult.

Concurrent Medication:

Excluded:

* Corticosteroid treatment (except replacement therapy or patients in Group B).
* Ganciclovir.
* Zidovudine (AZT).
* Investigational agents including antiretroviral agents (didanosine (ddI), dideoxycytidine (ddC), etc.).

Drugs likely to have anti-pneumocystis effect such as:

* Sulfonamides.
* Pentamidine.
* Dapsone.
* Trimethoprim.
* Other DHFR inhibitors.
* Primaquine.
* Clindamycin.
* Sulfonylureas.

Patients with the following are excluded:

* Judged by the investigator to be in impending respiratory failure.
* Prior therapy for this episode of PCP or treatment within 4 weeks of entry for a prior episode of PCP.
* Unable to or refuse to discontinue zidovudine, ganciclovir, or other antiretroviral agents during the 21 day treatment period.
* Unable to take medication orally or unwilling or unable to take study medication with food.
* Significant psychosis or emotional disorder such that, in the investigator's opinion, the patient would not be compliant with the study protocol.
* Prior documented glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Prior history of life-threatening toxicity to SMX/TMP such as severe rash or Stevens-Johnson syndrome.

Prior Medication:

Excluded:

* Prior therapy for this episode of Pneumocystis carinii pneumonia (PCP) or treatment within 4 weeks for a prior episode of PCP.
* Blood transfusions.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Primary Completion 1992-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hughes WT, Study Chair
Locations (38):
- United States (27):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Foundation Hosp, Harbor City, California
  - USC, Los Angeles, California
  - Dr Richard Meyer, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Infectious Disease Med Group, Oakland, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Dr Marcus Conant, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Dr Winkler Weinberg, Roswell, Georgia
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Natl Inst of Allergy & Infect Dis / Cln Ctr, Bethesda, Maryland
  - Washington Univ School of Medicine, St Louis, Missouri
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Good Samaritan Hosp, Portland, Oregon
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - The Regional Medical Ctr, Memphis, Memphis, Tennessee
  - Plaza Med Ctr, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
- CHU Saint Pierre, Brussels, Belgium
- Canada (3):
  - Dr Julio S G Montaner, Vancouver, British Columbia
  - Wellesley Hosp, Toronto, Ontario
  - Montreal Gen Hosp, Montreal, Quebec
- Hopital Bichat - Claude Bernard, Paris, France
- Germany (2):
  - August-Viktoria-Krankenhaus Chefarst derII Inneren Abteilung, Berlin
  - Universitat Munchen / Medizinische Poliklinik, Munich
- Natac Med Centre, Amsterdam, Netherlands
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico
- United Kingdom (2):
  - Kobler Centre / Saint Stephen's Hosp, London
  - Saint Mary's Hosp, London

REFERENCES:
- [Background] Hughes W, et al. Comparison of 566C80 & trimethoprim-sulfamethoxazole (TMP-SMZ) for the treatment of P. carinii pneumonitis (PCP). An International Multicenter, CCTG & ACTG Collaboration. Int Conf AIDS. 1992 Jul 19-24;8(1):We48 (abstract no WeB 1019)
- [Background] Hughes W, Leoung G, Kramer F, Bozzette SA, Safrin S, Frame P, Clumeck N, Masur H, Lancaster D, Chan C, et al. Comparison of atovaquone (566C80) with trimethoprim-sulfamethoxazole to treat Pneumocystis carinii pneumonia in patients with AIDS. N Engl J Med. 1993 May 27;328(21):1521-7. doi: 10.1056/NEJM199305273282103. PMID 8479489